CLINICAL TRIAL: NCT04044534
Title: Intranasal Insulin for Treating Posttraumatic Stress Disorder
Brief Title: Intranasal Insulin for Posttraumatic Stress Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gihyun Yoon, MD, Principal Investigator, VA Connecticut Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GY0005
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: PTSD
Keywords: Intranasal insulin; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal insulin (Experimental): Subjects in this arm will receive 40 IU of intranasal insulin twice a day (80 IU per day).
  Interventions: Drug: Intranasal insulin
- Placebo (Experimental): Subjects in this arm will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal insulin — Subjects in this arm will receive intranasal insulin (80 IU per day).
  Arms: Intranasal insulin
Drug: Placebo — Subjects in this arm will receive placebo.
  Arms: Placebo

SUMMARY:
To evaluate if intranasal insulin is effective in reducing PTSD symptoms.

DETAILED DESCRIPTION:
The current proposal aims to study the pharmacotherapeutic effects of intranasal insulin on PTSD symptoms and inhibition of amygdala hyperactivation in subjects with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21-65 years old
* Current PTSD
* Able to provide written informed consent

Exclusion Criteria:

* Unstable medical condition, clinically determined by a physician
* Diabetes requiring insulin or oral hypoglycemic agents
* Moderate-severe traumatic brain injury
* Current psychotic disorder, bipolar disorder, cognitive disorder in the past 12 months
* Current substance use disorders (except alcohol, tobacco, or cannabis) in the past 3 months
* Changes in doses of psychotropic medications in the past 4 weeks
* Initiation of individual therapy or counseling in the past 4 weeks
* Imminent suicidal or homicidal risk
* Contraindication to Insulin
* History of claustrophobia
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI safety screening questionnaire

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder (PTSD) symptoms as measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | 1 week
  The five-point CAPS-5 consists of 20 PTSD symptoms rated on a 0-4 scale (total range: 0-80) as follows: (1) 5 Intrusion symptoms (0-20), (2) 2 Avoidance symptoms (0-8), (3) 7 Cognitions and mood symptoms (0-28), and (4) 6 Arousal and reactivity symptoms (0-24). Higher scores represent a worse outcome (i.e., more PTSD symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Gihyun Yoon, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States